CLINICAL TRIAL: NCT00354263
Title: IMP321 Phase I Study of Four Increasing Doses (3, 10, 30 and 100 µg) of a New Immunostimulatory Factor (IMP321) Given Alone or as an Adjuvant to a Reference Flu Antigen in Healthy Young Male Volunteers
Brief Title: Phase I Study of IMP321 Given Alone or as an Adjuvant to a Reference Flu Antigen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immutep S.A.S. (Industry)
Collaborators: SGS Aster-Cephac (CRO) (Unknown)
Responsible Party: F. Triebel, Chief Medical Officer, Immutep S.A.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P001; Aster-P020255
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Healthy
Keywords: Healthy male volunteers; IMP321; Adjuvant; Monotherapy; Pharmacokinetics/Pharmacodynamics
MeSH Terms: interventions — soluble LAG-3 protein, human; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): PBS injected alone in step 1 or mixed with Aggripal in step 2
  Interventions: Biological: saline
- B (Experimental)
  Interventions: Biological: IMP321

INTERVENTIONS:
Biological: IMP321 — This study is a single centre, single blind, placebo (step 1) or reference (step 2) randomised study. Healthy young male volunteers will receive single ascending dose of IMP321 in each step (4 doses tested: 3, 10, 30 and 100 µg). In step 1, IMP321 will be given alone and tested versus placebo (physiological saline). In step 2, the association IMP321 + Agrippal (commercially available flu vaccine) will be tested versus Agrippal alone.
  Other Names: hLAG-3Ig; CD223; LAG-3
  Arms: B
Biological: saline — saline injected alone in step 1 or mixed with Aggripal in step 2
  Arms: A

SUMMARY:
This study is a single centre, single blind, placebo (step 1) or reference (step 2) randomised study. Healthy young male volunteers will receive single ascending dose of IMP321 in each step (4 doses tested: 3, 10, 30 and 100 µg). In step 1, IMP321 will be given alone and tested versus placebo (physiological saline). In step 2, the association IMP321 + Agrippal (commercially available flu vaccine) will be tested versus Agrippal alone.

DETAILED DESCRIPTION:
This study is divided in two steps:

Step 1 (20 volunteers): IMP321 will be given alone and tested versus placebo (physiological saline)

In this first step, 4 group doses (of four subjects each) will be evaluated versus a placebo group of 4 subjects:

* Group IMP321 alone at 3 µg,
* Group IMP321 alone at 10 µg,
* Group IMP321 alone at 30 µg,
* Group IMP321 alone at 100 µg.

In order to complete these groups, four successive cohorts of volunteers will be studied:

Cohort A will correspond to the dose 3 µg and will include:

* 4 subjects treated by IMP321 3 µg alone
* 1 subject treated by placebo

If the tolerability of this cohort is acceptable, the following cohort will be done.

Cohort B will correspond to the dose 10 µg and will include:

* 4 subjects treated by IMP321 10 µg alone
* 1 subject treated by placebo

If the tolerability of this cohort is acceptable, the following cohort will be dose.

Cohort C will correspond to the dose 30 µg and will include:

* 4 subjects treated by IMP321 30 µg alone
* 1 subject treated by placebo

If the tolerability of this cohort is acceptable, the following cohort will be done.

Cohort D will correspond to the dose 100 µg and will include:

* 4 subjects treated by IMP321 100 µg alone
* 1 subject treated by placebo

Step 2 (40 volunteers): The association IMP321 + Agrippal will be tested versus the Agrippal alone.

In this second step, 4 group doses (of eight subjects each) will be evaluated versus a reference group (Agrippal + physiological saline) of 8 subjects:

* Group Agrippal + 3 µg of IMP321,
* Group Agrippal + 10 µg of IMP321,
* Group Agrippal + 30 µg of IMP321,
* Group Agrippal + 100 µg of IMP321.

In order to complete these groups, four successive cohorts of volunteers will be studied.

Cohort A will correspond to the dose 3 µg of IMP321 and will include:

* 8 subjects treated by Agrippal + IMP321 3 µg
* 2 subjects treated by Agrippal + physiological saline

If the tolerability of this cohort is acceptable, the following cohort will be done.

Cohort B will correspond to the dose 10 µg of IMP321 and will include:

* 8 subjects treated by Agrippal + IMP321 10 µg
* 2 subjects treated by Agrippal + physiological saline

If the tolerability of this cohort is acceptable, the following cohort will be done.

Cohort C will correspond to the dose 30 µg of IMP321 and will include:

* 8 subjects treated by Agrippal + IMP321 30 µg
* 2 subjects treated by Agrippal + physiological saline

If the tolerability of this cohort is acceptable, the following cohort will be done.

Cohort D will correspond to the dose 100 µg of IMP321 and will include:

* 8 subjects treated by Agrippal + IMP321 100 µg
* 2 subjects treated by Agrippal + physiological saline.

This study will be a single centre, single blind, placebo (step 1) or reference (step 2) randomised study.

Healthy young male volunteers will receive single ascending dose of IMP321 in each step. Treatments will be administered as a subcutaneous injection on the mornings of Day 1. The injection will be done subcutaneously (s.c.) in the deltoid area of the non dominant arm.

The pharmacokinetic analysis will be performed by IMP321-specific ELISA testing of the samples collected from the 4 volunteers receiving 100 µg IMP321 alone. Blood samples will be taken on the morning of Day 1 before dosing then at 0.5, 1, 4, 24 and 48 h after dosing.

Blood samples (for T cell assays) and serum samples (for hLAG-3Ig- and HA-specific antibody detection by ELISA) will be taken on the morning of Days 1, 29 and 57.

Monitoring for the occurrence of adverse events (AE), changes in physical examination, vital signs (blood pressure, pulse rate, respiration), electrocardiograms (ECG) and clinical laboratory tests (biochemistry, haematology, urinalysis) will be performed before and after each dose of the study drug to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* able to give a written informed consent ;
* healthy male volunteers aged between 18 and 40 years;
* with body mass index (weight/height²) in the range 18 to 30 kg/m²;
* registered with the French Social Security in agreement with the French Law (Huriet Law : N° 88.1138 - 20.12.88) on biomedical experimentation;
* able to comply with protocol requirements, including blood and urine sample collections as defined in the protocol;
* not flu vaccination in the last two years.

Exclusion Criteria:

* who on direct questioning and physical examination have evidence of any clinically significant acute or chronic disease, including known or suspected HIV, HBV and HCV infection ;
* with any clinically significant abnormality following review of pre-study laboratory tests and full physical examination ;
* who have received any experimental drug within the exclusion period defined in the National Register for Healthy Volunteers of the French Ministry of Health ;
* who forfeit their freedom by administrative or legal award or who were under guardianship ;
* unwilling to give their informed consent ;
* who present a positive laboratory test for Hepatitis B surface antigen (HbsAg), HBc antibodies, HIV 1 and 2 antibodies and HCV antibodies ;
* who have a history of allergy or intolerance to the study drug ;
* who had a history of serious allergy, asthma, allergic skin rash or sensitivity to any drug ;
* who are known or suspected alcohol or drug abusers ;
* who present a positive laboratory test for urine drug screening (opiates, barbiturates, amphetamine, cannabis) ;
* who undergo surgery or have donated blood within 1 month prior to the start of the study ;
* who have taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 1 week prior to the first dose administration ;
* who receive any drug known to affect hepatic metabolism like cimetidine, ketoconazole, fluconazole, itraconazole, phenytoin, rifampicin, rifabutin within 1 month prior to the first dose administration ;
* who receive any drug known to affect renal tubular secretion like probenecid, beta-lactam antibiotics within 2 weeks prior to the first dose administration ;
* who present any clinical condition or prior therapy which, in the opinion of the investigator, made the subject unsuitable for the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2005-09 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To evaluate clinical and laboratory safety and tolerability profiles | 6 weeks

SECONDARY OUTCOMES:
To determine T cell response induction efficacy | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Didier Chassard, M.D., Principal Investigator — Aster-Cephac
Locations (1):
- SGS Aster-Cephac, Paris, France

REFERENCES:
- See also: Sponsor's website — http://www.immutep.com